CLINICAL TRIAL: NCT06121544
Title: The Swedish BioFINDER - Preclinical AD Study
Status: Recruiting | Type: Observational
Sponsor: Skane University Hospital (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Erik Stomrud, M.D., PhD, Skane University Hospital
Other Study IDs: SAIS
Record Dates: First submitted 2023-11-02; First posted 2023-11-08 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Mild Dementia
Keywords: Preclinical Alzheimer, early diagnosis, biomarkers, plasma, CSF, PET
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, cerebrospinal fluid (CSF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cognitively unimpaired individuals with preclinical Alzheimer's disease: 75% of the recruited population will be cognitively unimpaired individuals with preclinical Alzheimer's disease.
  Interventions: Diagnostic Test: Plasma tau; Diagnostic Test: Plasma Ab42/Ab40; Diagnostic Test: Flutemetamol F18 Injection; Diagnostic Test: [18F]-RO6958948 Injection; Diagnostic Test: Magnetic resonance imaging (MRI)
- Cognitively unimpaired individuals without preclinical Alzheimer's disease.: 25% of the recruited population will be cognitively unimpaired individuals without preclinical Alzheimer's disease.
  Interventions: Diagnostic Test: Plasma tau; Diagnostic Test: Plasma Ab42/Ab40; Diagnostic Test: Flutemetamol F18 Injection; Diagnostic Test: [18F]-RO6958948 Injection; Diagnostic Test: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Plasma tau — Plasma levels of different p-tau and np-tau species
Diagnostic Test: Plasma Ab42/Ab40 — Plasma levels of Ab42/Ab40 ratio
Diagnostic Test: Flutemetamol F18 Injection — Positron emission tomography (PET) imaging of amyloid-β plaques
Diagnostic Test: [18F]-RO6958948 Injection — PET imaging of Tau aggregates
Diagnostic Test: Magnetic resonance imaging (MRI) — Different MRI sequences relevant for brain imaging

SUMMARY:
This research study aims to examine biomarkers of Alzheimer's disease (AD) as early as possible which could potentially be a screening tool for the general population. This observational study will take place at the Skåne University Hospital in Sweden. The study will enroll up to 600 cognitively healthy subjects aged 50 to 80 years with 3/4 having preclinical Alzheimer's disease. Recruitment and enrollment will be ongoing for 2-3 years, and subject participation will be lasting approximately 4 years. Disclosure of AD risk assessments will be an optional procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50-80
2. Individuals aged 50-60 require at least one of the following risk factors for AD:

   1. Known APOE-E4 carrier
   2. Known 1st degree family history of dementia or severe memory loss with onset prior to 75.
   3. Known amyloid brain pathology by either CSF or PET scan.
3. Mini-Mental State Examination (MMSE) ≥26 (aged >65); MMSE ≥27 (aged 50-65).
4. Score of 12 or above on the Montreal Cognitive Assessment (MoCA) telephone version.
5. Speaks and understands Swedish to the extent that an interpreter is not necessary to fully understand the study information and cognitive tests.

6a. Preclinical AD subgroup (n=450): Amyloid pathology according to CSF AD biomarkers and Aβ-PET scans.

6b. Non-Preclinical AD subgroup (n=150): No sign of preclinical AD using CSF AD biomarkers or Aβ-PET scans.

Exclusion Criteria:

1. Fulfils the criteria for minor or major neurocognitive disorder according to The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
2. History of significant brain injury or other known neurologic disease or insult, resulting in lasting cognitive sequelae that would confound the assessment and staging of potential neurodegenerative disease.
3. Major depression, bipolar disorder, or recurrent psychotic disorders within the past year.
4. History of alcohol and/or substance abuse or dependence within the past year.
5. Significant unstable systemic illness or organ failure, such as terminal cancer, that makes it difficult to participate in the study.
6. Refusing or unable to complete baseline cognitive and biomarker assessments (i.e., cognitive testing, blood draw, MRI and PET).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cognitively unimpaired individuals (50-80 y) Step 1. Cognitively normal individuals will be screened using plasma p-tau217 (Eli Lilly-developed MSD method).
  Step 2. CSF AD biomarkers will be done in a subpopulation including all plasma p-tau217 positive individuals and randomly selected individuals with normal p-tau217 (matching 9:1).
  Step 3. Amyloid PET imaging.
  450 individuals with positive AD biomarkers and 150 with normal AD biomarkers will be enrolled into longitudinal study.
  FOLLOW-UP FOR 4 YEARS: Cognitive testing and blood draws will be conducted at baseline and 12, 24, 36 and 48 months. CSF collection, MRI, amyloid PET and tau PET will be conducted at baseline, and 24 and 48 months.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for 4 years after baseline.
  Rate of cognitive decline as measured by traditional cognitive and behavioral assessments including The Preclinical Alzheimer Cognitive Composite (PACC)
Change in cognitive function - digital assessment | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for 4 years after baseline.
  Rate of cognitive decline as measured by digital cognitive assessments

SECONDARY OUTCOMES:
Rate of change in plasma biomarkers | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every year for 4 years after baseline.
Rate of change in CSF biomarkers | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every two years for 4 years after baseline.
Rate of change in amyloid PET | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every two years for 4 years after baseline.
Rate of change in tau PET | Time zero equals the baseline visit. All subjects will subsequently attend follow-up visits every two years for 4 years after baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within one year after study completion